CLINICAL TRIAL: NCT02571608
Title: ContinuAtioN of meTformin to Improve And KEep Peri-operative Glycemic Control: A Randomized, Double-Blind, Placebo-Controlled Pilot Study.
Brief Title: Continuation of Metformin to Improve And Keep Peri-operative Glycemic Control
Acronym: CANTAKE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-152
Record Dates: First submitted 2015-09-29; First posted 2015-10-08 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Type 2 diabetes mellitus, Metformin, peri-operative
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Active Comparator): Metformin, dosage same as the patient's regular dosage
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — The study intervention involves Type II Diabetes Mellitus patient self-administered metformin vs. placebo according to regular dosing schedule and randomization. Both placebo and active drug will be over-encapsulated by pharmacy so that they will be indistinguishable to the personnel involved in the study.
  Other Names: Group A
  Arms: Metformin
Drug: Placebo — The study intervention involves Type II Diabetes Mellitus patient self-administered metformin vs. placebo according to regular dosing schedule and randomization. Both placebo and active drug will be over-encapsulated by pharmacy so that they will be indistinguishable to the personnel involved in the study.
  Other Names: Group B
  Arms: Placebo

SUMMARY:
Type II Diabetes Mellitus patients having surgery who adhere to their regular scheduled metformin dosing and take this medication on the morning of surgery will have better glycemic control peri-operatively and potentially suffer less morbidity compared to individuals taking a placebo.

DETAILED DESCRIPTION:
Peri-operative hyperglycemia has been linked to numerous negative adverse consequences, including wound infection, impaired wound healing, endothelial dysfunction, neurocognitive dysfunction, sepsis, prolonged hospital stay and increased mortality. This has been shown in numerous studies as outlined in our detailed research proposal. The peri-operative period includes a timeframe ranging from 12 to 72 hours around the time of surgery according to definition. Our study is examining glycemic control in the peri-operative period which we are defining as approximately 48 hours around the time of surgery. The majority of the patients with type II diabetes take oral medications, such as metformin, to control their blood sugar. These patients have historically held their doses on the day of the surgery to avoid possible low blood sugar and lactic acidosis while fasting. However, numerous recent studies have shown that individuals who are fasting without renal, heart and liver failure are safe to take metformin. The most recent guidelines from the American diabetes association suggest that patients should take their dose of metformin on the day of surgery. Despite these recommendations most anesthesiologists continue to withhold metformin on the day of surgery, as no studies exist to show the benefit of continuing metformin. If we are able to show that patients taken metformin have better glycemic control during this time we can extrapolate that result mean they may have a lower incidence of the consequences linked to poor glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 - 75, using metformin for control of Type II Diabetes mellitus, American Society of Anesthesiologists(ASA) I, II and III, informed consent, surgery in which less than 1000 mL of blood loss is expected.

Exclusion Criteria:

* renal failure, liver failure, Congestive heart failure (CHF), previous episodes of hypoglycemia, conditions which mask symptoms of hypoglycemia (autonomic neuropathy or chronic high dose beta-blocker usage), low capillary blood sugar (CBG) (≤4.0 mmol/L) at pre-operative appointment date, same day surgery, any patient who received contrast dye within 2 days of the planned surgery or requires intra-operative contrast dye and same day surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | One year
  This will be documented as total number of individuals recruited and randomized in the study.

SECONDARY OUTCOMES:
Glycemic control | Baseline, Intra-op, 1, 6, 12, 24 and 48 hours post-op
  Mean CBG score difference between 2 groups
Wound infection | At follow up visit with surgeon at approx. 6 weeks post-surgery
  Wound infection present at follow-up visit
Length of Hospital Stay | One year
  Mean length of stay for all patients

CONTACTS AND LOCATIONS:
Overall Officials: James Paul, MD, FRCPC, Principal Investigator — McMaster University; Russell Brown, MDMC, PhD, FRCPC, Principal Investigator — McMaster University